CLINICAL TRIAL: NCT05087719
Title: Effects of Proprioceptive Activities on Hand Function in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/20/0208
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Proprioceptive Disorders
Keywords: graphesthesia; stereognosis; stroke
MeSH Terms: conditions — Stroke; Somatosensory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The patients in the experimental group will get the hot pack initially for 15 minutes .Then for proprioception training of graphesthesia for 15 mints, therapist repeatedly draw some letter, figures, digit, shapes ,alphabets on the palm of hand/digits of patient.For Stereognosis therapist command the patient to close his or her eyes, then on affected hand put some different kinds of objects and shapes then ask the patient to identify that object, the object might be of any kind like a key, rubber a block or a coin etc. Total time for stereognosis was 15 minutes. For motor training patients were guided by the therapist to use his or her affected hand more. Then patient practiced some task like drawing writing his or her name, folding the towel or a paper, eating something with different speed, picking small objects like nails and put them in to small boxes, organize the cards etc. This training session required 15 minutes.
  Interventions: Combination Product: experimental group
- conventional treatment (Active Comparator): baseline treatment of hot pack for 15 minutes will be given.The patients in this group will get muscle strengthening exercise of the hand, Range of motion, and stretching of the hand muscles, 3 sets of 8 repetitions were given to the patient, gap of 2 minutes will be given between regimes. For 20 minutes this session will be given to patient by the therapist.
  Interventions: Combination Product: conventional treatment

INTERVENTIONS:
Combination Product: experimental group — patients will receive the hot pack initially for 15 minutes .Then for proprioception training of graphesthesia for 15 mints,stereognosis will be of 15 minutes. For motor training patients will practice 15 mints motor tasks
  Arms: experimental group
Combination Product: conventional treatment — patients will receive the baseline treatment of hot pack for 15 minutes. The patients in this group will get muscle strengthening exercise of the hand, Range of motion, and stretching of the hand muscles, 3 sets of 8 repetitions were given to the patient, gap of 2 minutes will be given between regimes. For 20 minutes this session will be given to patient by the therapist.
  Arms: conventional treatment

SUMMARY:
To determine effects of proprioceptive activities on hand function in chronic stroke patients

DETAILED DESCRIPTION:
Stroke is causing the long term disability worldwide. The patient in the chronic phase of stroke may suffer from long term hand disability along with both motor and sensory dysfunction. That causes hindrance in performing the ADLs. As the hand is the important organ performing major functions of daily living .So the early restoration of the motor as well as sensory function is necessary.

The motive of this study IS to determine effects of proprioceptive activities on hand function in chronic stroke patients. Total 40 chronic stroke patients will be included in the study. They will be randomly allocated in two groups by lottery method that fulfills the inclusion criteria of the study. In group A patients will be recruited and proprioceptive activities will be given to the affected hand for 3 days /week for 2 months. On the other hand in group B conventional therapy will be given for 3 days /week for 2 months. In sensory training graphesthesia and stereognosis will be checked by modified subtest of sensory integration praxis test and Byl-Cheney-Boczai Sensory Discriminator Test respectively. The motor task will be assessed by the wolf motor test. As a baseline treatment hot pack for 15 min will be given to both of the groups

ELIGIBILITY:
Inclusion Criteria:

* Either right or left sided hemiplegic patients post stroke 6 months to 4 years
* Can partially open and close hand and able to elevate arm to at least 60 degrees and bend to 45-60 degree against gravity.

Exclusion Criteria:

* Patient with TBI, neuromuscular degenerative diseases, diabetes, heart disease, fracture of hand ,.muscular skeletal injuries of hand or birth deformities of hand
* Patients having any known or diagnosed psychological condition or unable to follow the command for exercise.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
wolf motor assessment scale | 15 minutes
  The scale was categorized from 0-5.0 represents that UE doesn't attempt tested.1 represents that the UE being tested does not participate functionally.2 represents that UE does movements minor readjustment or change in position, but requires assistance.3 represents UE does movement but movements is effected to certain degree by synergy or performance gradually or with effort.4 represents that movement was close to normal slight slower lack accuracy.5 represents that movement seems to be accurate
Byl-Cheney-Boczai Sensory Discriminator Test | 15 minutes
  For the stereognosis
Graphesthesia (modified sub test of sensory integration praxis test) | 15 minutes
  to assess Graphesthesia

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CY, Fu T, Lin KC, Feng CT, Hsieh KP, Yu HW, Lin CH, Hsieh CJ, Ota H. Assessing the streamlined Wolf motor function test as an outcome measure for stroke rehabilitation. Neurorehabil Neural Repair. 2011 Feb;25(2):194-9. doi: 10.1177/1545968310381249. Epub 2010 Oct 14. PMID 20947494
- [Background] Turville ML, Cahill LS, Matyas TA, Blennerhassett JM, Carey LM. The effectiveness of somatosensory retraining for improving sensory function in the arm following stroke: a systematic review. Clin Rehabil. 2019 May;33(5):834-846. doi: 10.1177/0269215519829795. Epub 2019 Feb 25. PMID 30798643
- [Background] Hatem SM, Saussez G, Della Faille M, Prist V, Zhang X, Dispa D, Bleyenheuft Y. Rehabilitation of Motor Function after Stroke: A Multiple Systematic Review Focused on Techniques to Stimulate Upper Extremity Recovery. Front Hum Neurosci. 2016 Sep 13;10:442. doi: 10.3389/fnhum.2016.00442. eCollection 2016. PMID 27679565